CLINICAL TRIAL: NCT04556838
Title: A Phase 2a, Double-Masked, Randomized, Vehicle-controlled Trial Evaluating the Safety and Efficacy Activity of 1% and 5% VVN001 Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: Study of VVN001 Ophthalmic Solution in Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VivaVision Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVN001-CS-201
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Double-masked parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VVN001, 1% (Experimental): VVN001, 1% ophthalmic solution
  Interventions: Drug: VVN001 Ophthalmic Solution 1%
- VVN001, 5% (Experimental): VVN001, 5% ophthalmic solution
  Interventions: Drug: VVN001 Ophthalmic Solution 5%
- Vehicle (Placebo Comparator): VVN001 Ophthalmic Solution Placebo
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: VVN001 Ophthalmic Solution 1% — VVN001 Ophthalmic Solution 1%
  Arms: VVN001, 1%
Drug: VVN001 Ophthalmic Solution 5% — VVN001 Ophthalmic Solution 5%
  Arms: VVN001, 5%
Drug: Vehicle — VVN001 Ophthalmic Solution Vehicle
  Arms: Vehicle

SUMMARY:
This is a Phase 2a, multi-center, double-masked, randomized, vehicle-controlled, parallel-group study designed to evaluate the safety and tolerability and to explore the efficacy activity of VVN001 ophthalmic solution versus vehicle in subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to any study-related procedures .
* Are 18 years of age or older.
* Are willing and able to follow instructions and willing to be present for the required study visits for the duration of the study.
* Have a best corrected visual acuity (BCVA), using corrective lenses if necessary, in the qualifying eye(s) of +0.7 or better as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) at the screening visit and randomization visit.
* Have a history of dry eye disease in both eyes
* Are currently using artificial tears and have been using within 30 days of the screening visit.
* Have an Eye dryness score ≥40 at Visit 1 and ≥35 at Visit 2, one score for both eyes (0-100 point VAS)
* Have ongoing dry eye disease in the same eye or both eyes, as defined by all of the following criteria in the study eye and the same eye at Visit 1 and Visit 2:
* Inferior CFS (iCFS) score of ≥2 (NEI; 0-4 scale; using 0.5 unit increments)
* Have a Schirmer score (without anesthesia) of ≥1 and ≤7 mm/5 min.

Exclusion Criteria:

* Have a known hypersensitivity or contraindication to the IP or components of IP.
* Have a Schirmer score (without anesthesia) of <1 or >7 mm/5 min in the study eye.
* Have history of uncontrolled glaucoma, IOP over 21 mmHg in either eye at the screening visit or are being treated with eye drops for glaucoma in the study eye. Or the subject has had laser or surgery for glaucoma in the study eye within 90 days of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lexitas, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tauber J, Evans D, Segal B, Li XY, Shen W, Lu C, Novack GD; VVN001-CS201 Study Group. A phase 2a, double-masked, randomized, vehicle-controlled trial of VVN001 in subjects with dry eye disease. Ocul Surf. 2023 Apr;28:18-24. doi: 10.1016/j.jtos.2022.12.007. Epub 2022 Dec 29. PMID 36586669

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VVN001, 1% | VVN001, 5% | Vehicle
Started | 57 | 56 | 56
Completed | 53 | 53 | 51
Not Completed | 4 | 3 | 5
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Subject travel | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VVN001, 1% | VVN001, 5% | Vehicle | Total
Number analyzed (Participants) | 57 | 56 | 56 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 27 | 80
  >=65 years | 30 | 30 | 29 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (14.50) | 62.5 (11.68) | 62.6 (13.25) | 63.4 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 48 | 39 | 126
  Male | 18 | 8 | 17 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 16 | 12 | 42
  Not Hispanic or Latino | 43 | 40 | 44 | 127
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 1 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 13 | 10 | 29
  White | 43 | 41 | 41 | 125
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Inferior Corneal Fluorescein Staining [Mean (Standard Deviation); unit: units on a scale (0 none to 4 severe)] — Scale: 0 (none) to 4 (severe)
  units on a scale (0 none to 4 severe) | 2.45 (0.532) | 2.45 (0.537) | 2.44 (0.548) | 2.44 (0.536)
Eye Dryness Visual Analog Scale [Mean (Standard Deviation); unit: units on a scale] — Units on a scale: 0 (none) to 100 (severe)
  units on a scale | 66.5 (18.59) | 66.2 (15.43) | 64.9 (17.34) | 65.9 (17.09)
Total Corneal Fluorescein Staining [Mean (Standard Deviation); unit: units on a scale] — Scale: 0 (none) to 20 (severe)
  units on a scale | 6.64 (3.24) | 6.96 (2.97) | 6.18 (2.92) | 6.59 (3.04)
Regional corneal fluorescein staining [Mean (Standard Deviation); unit: units on a scale] — Scale: 0 (none) to 4 (severe)
  units on a scale | 2.45 (0.532) | 2.45 (0.537) | 2.44 (0.548) | 2.44 (0.536)

OUTCOME MEASURES:

1. Primary Outcome: Inferior Corneal Fluorescein Staining
Description: Mean change from baseline in Inferior corneal fluorescein staining. Negative number indicates improvement. Depending upon individual subject's baseline, this measure can range from -4 to +4.
Time Frame: Day 84
Population: Sample size reflects number of subjects evaluable at Day 84
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VVN001, 1% | VVN001, 5% | Vehicle
Number analyzed (Participants) | 54 | 53 | 51
score on a scale | -0.69 (0.77) | -.97 (0.81) | -0.72 (0.83)

2. Secondary Outcome: Total Corneal Fluorescein Staining
Description: Mean change from baseline in total corneal fluorescein staining Negative number indicates improvement. Depending upon individual subject's baseline, this measure can range from -20 to +20.
Time Frame: Day 84
Population: Sample size reflects number of subjects evaluable at Day 84
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VVN001, 1% | VVN001, 5% | Vehicle
Number analyzed (Participants) | 53 | 53 | 51
score on a scale | -1.75 (2.39) | -2.60 (3.25) | -0.79 (3.08)

3. Secondary Outcome: Regional Corneal Fluorescein Staining
Description: Mean change from baseline in temporal regional corneal fluorescein staining. Negative number indicates improvement. Depending upon individual subject's baseline, this measure can range from -4 to +4.
Time Frame: Day 84
Population: Sample size reflects number of subjects evaluable at Day 84
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VVN001, 1% | VVN001, 5% | Vehicle
Number analyzed (Participants) | 53 | 53 | 51
score on a scale | -0.20 (0.72) | -0.52 (0.87) | -0.11 (0.84)

4. Secondary Outcome: Eye Dryness
Description: Mean Change in Eye Dryness VAS. Negative number indicates improvement. Depending upon individual subject's baseline, this measure can range from -100 to +100..
Time Frame: Day 84
Population: Sample size reflects number of subjects evaluable at Day 84
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VVN001, 1% | VVN001, 5% | Vehicle
Number analyzed (Participants) | 53 | 54 | 51
score on a scale | -28.7 (27.4) | -22.2 (25.02) | -19.9 (29.0)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | VVN001, 1% | VVN001, 5% | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 3/56 | 6/57 | 2/56
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VVN001, 1% (N=56) | VVN001, 5% (N=57) | Vehicle (N=56)
Chalzion (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Instillation site pain (Eye disorders) | 3 (3) | 1 (2) | 2 (2)
Dysguesia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT04556838/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT04556838/SAP_001.pdf